CLINICAL TRIAL: NCT00545818
Title: An Open, Prospective, Randomized, Multi-center Study Comparing OsseoSpeed™ Implant 6 mm With OsseoSpeed™ Implant 11 mm in the Posterior Maxilla and Mandible. A 5-year Follow-up Study.
Brief Title: Study Comparing OsseoSpeed™ Implants of Two Different Lengths in the Upper and Lower Posterior Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-SHO-0001
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-1, Implant length 6 mm (Experimental): Subjects treated with OsseoSpeed™ implant, length: 6 mm
  Interventions: Device: OsseoSpeed™ length 6 mm
- Group-2, Implant length 11 mm (Other): Subjects treated with OsseoSpeed™ implant, length: 11 mm
  Interventions: Device: OsseoSpeed™ length 11 mm

INTERVENTIONS:
Device: OsseoSpeed™ length 6 mm — OsseoSpeed™ dental implant, length: 6 mm
  Arms: Group-1, Implant length 6 mm
Device: OsseoSpeed™ length 11 mm — OsseoSpeed™ dental implant, length: 11 mm
  Arms: Group-2, Implant length 11 mm

SUMMARY:
The purpose of this study is to see if OsseoSpeed™ implant 6 mm long is effective for rehabilitation of edentulism and if so, how it compares with OsseoSpeed™ implant 11 mm long. The primary hypothesis is that the alteration in bone level is equal in patients randomized to 6 mm as to patients randomized to 11 mm implants.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Aged 20-70 years at enrolment
* History of edentulism in the study area of at least four months
* Neighboring tooth/teeth to the planned bridge must have natural root(s)
* Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned bridge.
* Deemed by the investigator to have a bone height of at least 11 mm and a bone width of minimum 6 mm
* Deemed by the investigator as likely to present an initially stable implant situation

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, as judged by the investigator
* Earlier graft procedures in the study area
* Uncontrolled pathologic processes in the oral cavity
* Known or suspected current malignancy
* History of radiation therapy in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
* Uncontrolled diabetes mellitus
* Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
* Smoking more than 10 cigarettes/day
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
* Previous enrolment in the present study.
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech
* Simultaneous participation in another clinical study, or participation in a clinical study during the last 6 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2007-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Karin Lundgren, Study Director — Direktor Clinical Research, Dentsply Sirona Implants, Mölndal, SWEDEN
Locations (6):
- United States (2):
  - USC School of Dentistry, Los Angeles, California
  - The University of Iowa, College of Dentistry, Iowa City, Iowa
- School of Dental Science, University of Melbourne, Melbourne, Victoria, Australia
- Praktijk De Mondhoek, Apeldoorn, Netherlands
- Dept. of Parodontology, Göteborg University, Gothenburg, Sweden
- King's College London Dental Institute at Guy's King's and St Thomas' Hospitals, London, United Kingdom

REFERENCES:
- [Result] Gulje F, Abrahamsson I, Chen S, Stanford C, Zadeh H, Palmer R. Implants of 6 mm vs. 11 mm lengths in the posterior maxilla and mandible: a 1-year multicenter randomized controlled trial. Clin Oral Implants Res. 2013 Dec;24(12):1325-31. doi: 10.1111/clr.12001. Epub 2012 Sep 3. PMID 22938573
- [Result] Zadeh HH, Gulje F, Palmer PJ, Abrahamsson I, Chen S, Mahallati R, Stanford CM. Marginal bone level and survival of short and standard-length implants after 3 years: An Open Multi-Center Randomized Controlled Clinical Trial. Clin Oral Implants Res. 2018 Aug;29(8):894-906. doi: 10.1111/clr.13341. Epub 2018 Jul 12. PMID 30003598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 97 subjects were enrolled in the study (singed informed consent).Two of those subjects fulfilled exclusion criteria and were removed from the study population before randomization.
  As a consequence a total of 95 subjects were randomised (assigned to groups) and received study treatment.
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Started | 49; 108 Implants | 46; 101 Implants
Completed | 46; 98 Implants | 39; 86 Implants
Not Completed | 3; 10 Implants | 7; 15 Implants
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.39) | 54.1 (10.04) | 54.5 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 47
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: participants]
  Sweden | 3 | 2 | 5
  Netherlands | 17 | 16 | 33
  United States | 18 | 14 | 32
  United Kingdom | 7 | 8 | 15
  Australia | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Radiological Assessments of Marginal Bone Level Alteration
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant.
  Marginal Bone Level expressed in millimeters at the 5 year follow-up visit compared to values obtained at delivery of temporary restoration i.e. loading (baseline).
  Positive value = bone gain, Negative value = bone loss.
Time Frame: Evaluated from implant installation to 5 years follow-up after implant placement
Population: A total of 85 subjects (184 implants) completed the study. For a total of 10 implants (in 5 subjects) the quality of the radiographs were not sufficient for reading, giving a total of 80 subjects (174 implants) for the analysis of MBL change.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Number analyzed (Participants) | 44 | 36
Number analyzed (Implants) | 94 | 80
millimeter | 0.02 (0.52) | -0.18 (1.05)

2. Secondary Outcome: Overall Implant Survival
Description: Overall implant survival, measured on implant level
Time Frame: Evaluated 5 years after implant placement
Population: Group-1. A total of 49 subjects (108 positions) underwent surgery. Three positions were not implanted due to complications during surgery. Giving a total 105 implants installed.
  Group-2. A total of 46 subjects (101 positions) underwent surgery. Giving a total of 101 implants installed.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Number analyzed (Participants) | 49 | 46
Number analyzed (implants) | 105 | 101
implants | 101 | 100

3. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment BoP
Description: Condition of the periimplant mucosa by assessment of Bleeding on Probing (BoP). Presented as s count of implants that show presence of BoP.
Time Frame: Measured at the 5-year follow-up visit after loading
Population: A total of 85 subjects (184 implants) completed the 5-year follow-up visit. All included in the assessment of BoP.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Number analyzed (Participants) | 46 | 39
Number analyzed (implants) | 98 | 86
implants | 43 | 28

4. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of Change in PPD
Description: Condition of the periimplant mucosa by assessment of change in probing pocket depth (PPD).
  Change in pocket depth expressed in millimeters at the 5-year follow-up visit, compared to values obtained at delivery of permanent restoration, i.e. loading (baseline).
  Negative value = increased pocket depth.
Time Frame: Evaluated at implant loading and at the 5-year follow-up visit.
Population: A total of 85 subjects (184 implants) completed the 5-year follow-up visit. Group-1. For 3 subjects (7 implants) the radiographs were not possible to evaluate, giving a total of 43 subjects (91 implants) being available for evaluation of change in PPD.
  Group-2. All radiographs readable, giving 39 subjects (86 positions) for the evaluation.
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: implants
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Number analyzed (Participants) | 43 | 39
Number analyzed (implants) | 91 | 86
millimeters | -0.57 (0.92) | -1.11 (1.77)

5. Secondary Outcome: Presence of Plaque
Description: Presence of plaque was evaluated at four surfaces around each study position (mesial, facial, distal and lingual). Plaque was recorded as presence or absence of plaque by visual inspection.
  A study position was considered as bleeding "yes" if at least one of the four surfaces around the implant showed presence of bleeding on probing.
Time Frame: Evaluated at the 5-year follow-up visit after loading.
Population: A total of 85 subjects (184 implants) completed the 5-year follow-up visit. All included in the assessment of presence of plaque.
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Number analyzed (Participants) | 46 | 39
Number analyzed (implants) | 98 | 86
implants | 16 | 6

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group-1, Implant Length 6 mm | Group-2, Implant Length 11 mm
Serious Adverse Events (participants affected / at risk) | 8/49 | 5/46
Other Adverse Events (participants affected / at risk) | 13/49 | 12/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-1, Implant Length 6 mm (N=49) | Group-2, Implant Length 11 mm (N=46)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Osteopaenia, trauma - fractured toes (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insufficient renal function (30%) (Renal and urinary disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Undefined heart problems (Cardiac disorders) | 1 (1) | 0 (0)
Failure knee-prosthesis (Product Issues) | 1 (1) | 0 (0)
Hip function failure (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Gallbladder removed (Hepatobiliary disorders) | 1 (1) | 0 (0)
Right hip replacement, post-op infection (Infections and infestations) | 1 (1) | 0 (0)
Armpit abscess due to spider bite. (Infections and infestations) | 1 (1) | 0 (0)
Bilateral toe infection (Infections and infestations) | 1 (1) | 0 (0)
Liver cancer (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Broken pelvis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonitis - Non Hodgkin disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hip fracture due to car accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Eye cancer (basal cell carcinoma) (Eye disorders) | 0 (0) | 1 (2)
Squamous cell skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-1, Implant Length 6 mm (N=49) | Group-2, Implant Length 11 mm (N=46)
Study implant failure (Product Issues) | 5 (5) | 1 (1) — Study implant failure (including implant mobility, excessive bone loss around implant and, implant related pain)
Bridge screw loosening (Product Issues) | 5 (5) | 5 (10) — Loosening of the screw attaching the restoration (the bridge) to the implant abutment.
Abutment fracture (Product Issues) | 1 (4) | 3 (3) — Fracture of the abutment connecting the implant with the restoration
Fracture of temporary bridge (Product Issues) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less